CLINICAL TRIAL: NCT01031186
Title: A First Time in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of GSK356278 (PDE4 Inhibitor) in Healthy Volunteers
Brief Title: First Time in Human Study
Acronym: FTIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113324
Record Dates: First submitted 2009-11-05; First posted 2009-12-14 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: healthy male volunteers; GSK356278; first time in man; major depressive disorder
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depressive Disorder, Major | interventions — 5-(5-((2,4-dimethylthiazol-5-yl)methyl)-1,3,4-oxadiazol-2-yl)-1-ethyl-N-(tetrahydro-2H-pyran-4-yl)-1H-pyrazolo(3,4-b)pyridin-4-amine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1, Session 1 (Experimental): In Dosing Session 1, the subjects will be administered 0.5 mg GSK356278 and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 1, Session 2 (Experimental): In Dosing Session 2, the subjects will be administered GSK356278 (0.5 mg and 1.5 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 1, Session 3 (Experimental): In Dosing Session 3, the subjects will be administered GSK356278 (1.5 mg and 4 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 1, Session 4 (Experimental): In Dosing Session 4, the subjects will be administered GSK356278 (4 mg and 8 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 1, Session 5 (Experimental): In Dosing Session 5, the subjects will be administered GSK356278 8 mg and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 2, Session 1 (Experimental): In Dosing Session 1, the subjects will be administered 8 mg GSK356278 and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 2, Session 2 (Experimental): In Dosing Session 2, the subjects will be administered GSK356278 (8 mg and 16 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 2, Session 3 (Experimental): In Dosing Session 3, the subjects will be administered GSK356278 (16 mg and 30 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 2, Session 4 (Experimental): In Dosing Session 4, the subjects will be administered GSK356278 (30 mg and 50 mg) and placebo in a fasted state.
  Interventions: Drug: GSK356278; Drug: PLACEBO
- Cohort 2, Session 5 (Experimental): In Dosing Session 5, the subjects will be administered GSK356278 50 mg and placebo in a fasted state. The subjects will undergo food assessment session in Session 5 incase they experience nausea. In food assessment session, the subjects will receive a dose of GSK356278 after a standard breakfast.
  Interventions: Drug: GSK356278; Drug: PLACEBO

INTERVENTIONS:
Drug: GSK356278 — GSK356278
Drug: PLACEBO — PLACEBO

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of GSK356278 in male volunteers

DETAILED DESCRIPTION:
To evaluate the safety, tolerability and pharmacokinetics of single ascending doses of GSK356278 and may assess the effect of food on GSK356278 pharmacokinetics. They study will assess the compound's effect on nausea, emesis and alertness. Close monitoring of cardiovascular parameters will be included.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphate and bilirubin less than or equal to 1.5 times upper limit of normal.
* Healthy as determined by a responsible and experienced physician based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Males aged between 18 and 65 years inclusive at the time of signing the informed consent.
* Males must agree to appropriate forms of contraception from administration of first dose through to 3 months after taking the final dose.
* Body weight greater than or equal to 50 kg and BMI within the range of 18-29.9 m2 (inclusive)
* Capable of giving written informed consent.
* QTcB or QTcF less than 450 msec

Exclusion Criteria:

* A positive pre-study Hep B or positive Hep C result within 3 months of screening.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities
* A positive pre-study alcohol and drug screen
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units or average daily intake of greater than 3 units
* The subject has participated in a clinical trial and has received investigational product within the time period of 30 days prior to first dosing day (or 5 half-lives or twice the duration of the biological effect of the drug, whichever is longer)
* Exposure to more than 4 new chemical entities in the last 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose unless in the opinion of the investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medication or history of drug or other allergy that in the opinion of the investigator or medical monitor contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Unwillingness or inability to follow the procedures in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects who have asthma or a history of asthma.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco or nicotine containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose.
* History of any significant psychiatric illness.
* Any history of suicidal behaviour or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale in the last 6 months.
* History of presence of clinically significant cardiac arrhythmias or other clinically significant cardiac disease.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2010-04-07 (Actual); Study Completion 2010-04-07 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of single escalating oral doses of GSK356278 in healthy male volunteers | 72 hours

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of single escalating doses of GSK356278 in healthy male volunteers | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 113324 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113324?search=study&search_terms=113324#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113324 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register